CLINICAL TRIAL: NCT04566263
Title: Treatment of Intracranial Wide-neck Aneurysms Using Stent-assisted Coil Embolization with the Stryker Neuroform EZ and Neuroform Atlas Stent Systems
Brief Title: Treatment of Intracranial Wide-neck Aneurysms Using Stent-assisted Coil Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002.VAS.2017.D
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: the Neuroform EZ Stent System was initially developed by SMART Therapeutics (San Leandro, CA, USA), with FDA HDE approval in 2002. This Stent system was later acquired by Boston Scientific, and then later acquired by Stryker Inc., Neurovascular Division. The Stent system was initially named the "Neuroform Microdelivery Stent System", and now has been re-branded as the "Neuroform EZ Stent System",
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Successful embolization of intracranial aneurysms (Other): Successful embolization of intracranial aneurysms defined by angiographic occlusion of greater than or equal to 90% at 6 months.
  Interventions: Device: Neuroform EZ Stent System

INTERVENTIONS:
Device: Neuroform EZ Stent System — The Stryker Neuroform EZ Stent System is a self-expanding nitinol, compliant, open-cell design that can be deployed by a single operator. The Neuroform EZ Stent System is packaged sterile as a single unit with an introducer sheath and a detachable push wire.

SUMMARY:
This device was designed to assist in the stent-assisted coil embolization of intracranial aneurysms, specifically those that have a wide neck that would not otherwise maintain the coil embolization material within the aneurysm because of the wide opening at the base of the aneurysm. This device was designed to treat aneurysms that are: unruptured, wide-necked, intracranial, saccular aneurysms arising from a parent vessel ≥ 2 mm and ≤ 4.5 mm. Wide-necked was defined as having a neck > 4mm or dome-to-neck ratio < 2.

DETAILED DESCRIPTION:
This is a prospective study to investigate the efficacy of using stent-assistance for embolization of intracranial aneurysms with a wide neck (defined as > or = to 4mm, or with a dome to neck ratio of 2:1 or less). We plan to investigate successful embolization of intracranial aneurysms defined by angiographic occlusion of greater than or equal to 90% at 6 months. Patients will be followed for a minimum period of 2 years from the date of the procedure, with a planned total duration of 4 years of the study, including follow up time. Participants will be initially assessed and if included, will undergo procedure that includes use of the device. Afterwards, they will be scheduled for regular follow up at 2 weeks for clinical assessment, then again at 3 months for clinical assessment and MRA to investigate the stented region, then again at 6 months for clinical assessment and possible cerebral angiogram vs possible MRA, and then again at 1 year post-procedure, and then again at 2 years post-procedure. Patients may then follow up on an annual basis or every 2-3 years, depending on preference and any residual or recurrent aneurysm. A more specific timeline and treatment course is described below.

Patients will receive cerebral angiography for evaluation of their cerebral vasculature and aneurysm configuration to ensure that the parent vessel diameter is adequate and that the aneurysm is 4mm in size with a wide neck. In these cases, if it is determined that the patient will require additional vascular support in order to adequately embolize the aneurysm then the use of stent-assisted coil embolization may be offered to the patient.

Once enrolled, patients will undergo endovascular stent-assisted coil embolization of the aneurysm, and clinical outcomes will then be assessed. Data will be collected for analysis according to the primary and secondary outcome measures in addition to any deviations from the protocol or safety concerns as well

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old or older) with intracranial aneurysms with a wide neck (defined as > or = to 4mm, or with a dome to neck ratio of 2:1 or greater).

Exclusion Criteria:

* Small-necked aneurysms,
* Inability to tolerate anti-platelet medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Angiographic occlusion | 6 months
  Successful embolization of intracranial aneurysms defined by angiographic occlusion of greater than or equal to 90%

CONTACTS AND LOCATIONS:
Overall Officials: Bartley Mitchell, M.D., Principal Investigator — Methodist Brain and Spine Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No